CLINICAL TRIAL: NCT02681822
Title: Multi-center Imaging Genetics Studies in China
Acronym: CHIMGEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Tianjin Medical University Second Hospital (Other); Tianjin First Central Hospital (Other); Pingjin Hospital,Logistics University of Chinese People's Armed Police Forces (Unknown); School of Medical Imaging, Tianjin Medical University (Unknown); Tianjin Huanhu Hospital (Other); Beijing Hospital (Other Government); Chinese PLA General Hospital (Other); Beijing Tongren Hospital (Other); Xuanwu Hospital, Beijing (Other); Peking Union Medical College Hospital (Other); Beijing Normal University (Other); Chinese Academy of Sciences (Other Government); The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Inner Mongolia Medical College Hospital (Unknown); The First Hospital of Jilin University (Other); The Frist Hospital Of China Medical University (Unknown); The First Affiliated Hospital of Dalian Medical University (Other); RenJi Hospital (Other); Huashan Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Nanjing PLA General Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Xuzhou Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Shan dong Medical Imaging Research Institute (Unknown); Qilu Hospital of Shandong University (Other); Yantai Yuhuangding Hospital (Other); Henan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Tongji Hospital (Other); Wuhan University (Other); Xiangya Hospital of Central South University (Other); Central South University (Other); Guangdong Provincial People's Hospital (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); South China Normal University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Xijing Hospital (Other); Tang-Du Hospital (Other); LanZhou University (Other); West China Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); University of Electronic Science and Technology of China (Other); First Affiliated Hospital of Chongqing Medical University (Other); Southwest Hospital, China (Other); The University of Science and Technology of China (Other); Guangdong No.2 Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Chunshui Yu, Head of Department of Radiology and Tianjin Key Laboratory of Functional Imaging, Tianjin Medical University General Hospital
Other Study IDs: 81425013
Record Dates: First submitted 2016-02-07; First posted 2016-02-12 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer Disease; Schizophrenia; Major Depressive Disorders
Keywords: Genome-wide association studies; Environmental factors; Behavioral Assessment; Pathway analysis
MeSH Terms: conditions — Alzheimer Disease; Schizophrenia; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators retain the peripheral blood drawn from antecubital vein in order to acquire the genotype, whether the healthy young participants carry the risk allele of one specific gene or not. No matter what genotypes the participants own, no specific intervention measure will be done among the participants.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy young subjects: Healthy young Chinese Han subjects aged 18-30

SUMMARY:
To study the impact of genetic and environmental factors on high-level cognition associated neural circuits among healthy young Chinese Han subjects.

DETAILED DESCRIPTION:
The investigators plan to collect behavioral assessment and environmental factors data,peripheral blood sample, MRI brain images in more than 10,000 healthy young Chinese Han individuals in order to build the pathway from gene to high-level cognitive phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-30
* Chinese Han
* right-handed
* without history of neuropsychiatric disease
* no substance addiction
* smoking

Exclusion Criteria:

* younger or elder than 18-30 year-old
* other ethnics
* with history of neuropsychiatric disease
* with history of neuropsychiatric disease among first,second and third degree relatives

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young Chinese Han subjects age 18-30
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-11; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Brain structure and function measured by MRI scans | 2 years
  The participants will receive non-interventional multi-modal MRI scans, such as 3D-T1WI, DTI, DKI, ASL, REST-fmri, then the investigators can acquire the brain volume in region of interest, such as bilateral hippocampus.

SECONDARY OUTCOMES:
Childhood adversities as assessed by Childhood Trauma Questionnaire-Short Form (Chinese Version) | 2 years
  To investigate impact of the adversities in early life of participants on brain structure and function as well as the interaction effect of childhood adversities and genetic variations,such as 5-HTTLPR polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Chunshui Yu, PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the IPD with the member institutes or hospitals after the total completion of the investigation.

REFERENCES:
- [Background] Braskie MN, Jahanshad N, Stein JL, Barysheva M, McMahon KL, de Zubicaray GI, Martin NG, Wright MJ, Ringman JM, Toga AW, Thompson PM. Common Alzheimer's disease risk variant within the CLU gene affects white matter microstructure in young adults. J Neurosci. 2011 May 4;31(18):6764-70. doi: 10.1523/JNEUROSCI.5794-10.2011. PMID 21543606
- [Background] Corder EH, Saunders AM, Strittmatter WJ, Schmechel DE, Gaskell PC, Small GW, Roses AD, Haines JL, Pericak-Vance MA. Gene dose of apolipoprotein E type 4 allele and the risk of Alzheimer's disease in late onset families. Science. 1993 Aug 13;261(5123):921-3. doi: 10.1126/science.8346443.